CLINICAL TRIAL: NCT06446726
Title: Efficacy and Safety of Low-dose Radiation Combined With Neoadjuvant Chemotherapy and Immunotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Low-dose Radiation Combined With Neoadjuvant Immunochemotherapy for Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Bo Zhang, Principal investigator, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDRT-2025
Record Dates: First submitted 2024-05-16; First posted 2024-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; low-dose radiation; neoadjuvant immunochemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Radiotherapy; 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Intervention Model Description: Group 1 (10 patients): Patients received neoadjuvant low-dose radiotherapy (4 Gy/2 fractions) combined with a domestic PD-1 inhibitor (tislelizumab) and chemotherapy as neoadjuvant therapy.
  Group 2 (10 patients): Patients received neoadjuvant low-dose radiotherapy (6 Gy/3 fractions) combined with a domestic PD-1 inhibitor (tislelizumab) and chemotherapy as neoadjuvant therapy.
  Group 3 (10 patients): Patients received neoadjuvant low-dose radiotherapy (8 Gy/4 fractions) combined with a domestic PD-1 inhibitor (tislelizumab) and chemotherapy as neoadjuvant therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4Gy/2f group (Experimental): During the neoadjuvant treatment phase, patients will undergo two cycles of low-dose radiotherapy, combined with chemotherapy and immunotherapy, each cycle lasting 21 days. The specific treatment protocol is as follows:
  D1/2: Low-dose radiotherapy (4 Gy/2f) D3: Tislelizumab, fixed dose of 200 mg; Nab-paclitaxel 260 mg/m2; Cisplatin 75 mg/m2. The interval between radiotherapy and chemotherapy should not exceed 3 days. Drug infusions follow the sequence of tislelizumab → nab-paclitaxel → cisplatin/carboplatin, with at least a 30-minute interval between each infusion.
  At the end of the neoadjuvant treatment, patients will undergo surgical treatment 6-8 weeks after the last treatment session.
  Interventions: Drug: Tislelizumab; Radiation: Low-dose radiotherapy; Drug: Nab-paclitaxel; Drug: Cisplatin
- 6Gy/3f group (Experimental): During the neoadjuvant treatment phase, patients will undergo two cycles of low-dose radiotherapy, combined with chemotherapy and immunotherapy, each cycle lasting 21 days. The specific treatment protocol is as follows:
  D1/2/3: Low-dose radiotherapy (6 Gy/3f) D4: Tislelizumab, fixed dose of 200 mg; Nab-paclitaxel 260 mg/m2; Cisplatin 75 mg/m2. The interval between radiotherapy and chemotherapy should not exceed 3 days. Drug infusions follow the sequence of tislelizumab → nab-paclitaxel → cisplatin/carboplatin, with at least a 30-minute interval between each infusion.
  At the end of the neoadjuvant treatment, patients will undergo surgical treatment 6-8 weeks after the last treatment session.
  Interventions: Drug: Tislelizumab; Radiation: Low-dose radiotherapy; Drug: Nab-paclitaxel; Drug: Cisplatin
- 8Gy/4f group (Experimental): During the neoadjuvant treatment phase, patients will undergo two cycles of low-dose radiotherapy, combined with chemotherapy and immunotherapy, each cycle lasting 21 days. The specific treatment protocol is as follows:
  D1/2/3/4: Low-dose radiotherapy (8 Gy/4f) D5: Tislelizumab, fixed dose of 200 mg; Nab-paclitaxel 260 mg/m2; Cisplatin 75 mg/m2. The interval between radiotherapy and chemotherapy should not exceed 3 days. Drug infusions follow the sequence of tislelizumab → nab-paclitaxel → cisplatin/carboplatin, with at least a 30-minute interval between each infusion.
  At the end of the neoadjuvant treatment, patients will undergo surgical treatment 6-8 weeks after the last treatment session.
  Interventions: Drug: Tislelizumab; Radiation: Low-dose radiotherapy; Drug: Nab-paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Tislelizumab — Patients will undergo two cycles of immunotherapy, each cycle lasting 21 days. Day 3 and Day 24: Tislelizumab, fixed dose of 200 mg
  Other Names: Tislelizumab, fixed dose of 200 mg
Radiation: Low-dose radiotherapy — Patients will undergo two cycles of low-dose radiotherapy. Day 1/2 and Day 22/23: Low-dose radiotherapy (8 Gy/4f)
  Other Names: Low-dose radiotherapy (8 Gy/4f)
Drug: Nab-paclitaxel — Patients will undergo two cycles of chemotherapy. Day 3 and Day 24: Nab-paclitaxel 260 mg/m2
  Other Names: Nab-paclitaxel 260 mg/m2
Drug: Cisplatin — Patients will undergo two cycles of chemotherapy. Day 3 and Day 24: Cisplatin 75 mg/m2.
  Other Names: Cisplatin 75 mg/m2

SUMMARY:
This study aims to investigate the efficacy and safety of low-dose radiation combined with neoadjuvant chemotherapy and immunotherapy in the treatment of locally advanced thoracic esophageal squamous cell carcinoma. By reducing the radiation dose from 40 Gy in 20 fractions to 4 Gy in 2 fractions, the goal is to lessen the adverse reactions caused by radiotherapy. Additionally, the study explores whether low-dose radiation therapy can promote the cross-presentation of tumor-specific antigens and increase lymphocyte infiltration into the tumor site. Study also examines whether this approach can enhance tumor-specific immune responses, thereby potentially improving the efficacy of immune checkpoint inhibitors.

DETAILED DESCRIPTION:
According to 2020 GLOBOCAN data, esophageal cancer ranks fifth in incidence among all malignant tumors in China, with new cases reaching 324,000 and annual deaths at 301,000. These figures indicate a significant burden of esophageal cancer in China, accounting for 55% of esophageal cancer cases globally. Unlike in Western countries, most esophageal cancer patients in China have squamous cell carcinoma, and 40% are diagnosed at an advanced stage. Surgery is a key treatment for locally advanced esophageal cancer, but patients may achieve better clinical outcomes if they receive neoadjuvant therapy before surgery. However, the prognosis for these patients remains relatively poor. From 2009 to 2015, the overall 5-year relative survival rate for esophageal cancer was 21.4%, with local tumors at 46.7%, regional metastasis at 25.1%, and distant metastasis at only 4.8%.

In recent years, immunotherapy has shown significant survival benefits in patients with advanced esophageal cancer. Immuno-chemotherapy has now become the standard first-line treatment for advanced esophageal cancer. Currently, the introduction of immunotherapy as neoadjuvant treatment in locally advanced esophageal cancer is a highly regarded research area. Many studies are underway involving the combined application of neoadjuvant chemotherapy and immunotherapy, as well as neoadjuvant chemoradiotherapy and immunotherapy. Regarding safety, tislelizumab is similar to foreign similar drugs, mostly causing grade 1-2 adverse reactions, and is within a controllable range. Our center's previous research results have shown that tislelizumab can be used as a neoadjuvant immunotherapy drug for esophageal squamous cell carcinoma, with good perioperative safety.

It is worth noting that recent study reports indicate that the pathological complete response (PCR) rate of neoadjuvant chemotherapy combined with immunotherapy in small sample studies ranges from 17% to 22%, showing significant heterogeneity. Recently, Chinese scholars published a study in the international authoritative academic journal "Nature Medicine," indicating that using a PD-L1 antibody for immunotherapy combined with surgery, although the PCR rate was only 8%, the long-term survival effect was comparable to traditional chemoradiotherapy. This further proves that compared to traditional neoadjuvant chemoradiotherapy, neoadjuvant immunotherapy has broad development potential. However, the local control effects of immunotherapy alone or combined with chemotherapy are still unsatisfactory, which may affect the radical outcome of surgery and the long-term survival of patients. Therefore, combining more effective local treatment methods with immunotherapy is undoubtedly a more promising treatment option.

Low-dose radiotherapy (LDRT) is generally defined as a treatment not exceeding 2 Gy per session, totaling no more than 10 Gy, and is considered a non-ablative treatment [13]. The low toxicity of low-dose radiotherapy makes it a treatment option for those not suitable for body-targeted radiation therapy. Furthermore, although low-dose radiotherapy does not directly kill cancer cells, it can promote tumor regression by readjusting the tumor immune microenvironment.

Low-dose radiotherapy damages cell DNA, causing previously hidden or difficult-to-recognize tumor antigens to be exposed on the cell surface. This change promotes the cross-presentation of tumor-specific antigens, increases lymphocyte infiltration into the tumor site, enhances tumor-specific immune responses, and further improves the efficacy of immune checkpoint inhibitors. Preoperative immunotherapy can activate the patient's immune system, enabling it to recognize tumor antigens and establish immune memory. This allows the immune system to continue to function in immune surveillance after the surgical removal of the tumor. Currently, the main focus of clinical research is on how to maximize the synergistic effects between different treatment modalities to achieve the best survival outcomes for patients with locally advanced esophageal cancer while minimizing treatment side effects.

This study is a phase IIa clinical trial focusing on preliminary efficacy and safety. The study proposes a comprehensive treatment of neoadjuvant low-dose radiotherapy combined with chemotherapy and immunotherapy (chemoradiotherapy plus immunotherapy). By reducing the radiotherapy dose, the aim is to enhance local control efficacy while minimizing adverse reactions caused by the combined treatment regimen.

The plan involves neoadjuvant low-dose radiotherapy combined with chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma, with radiotherapy doses adjusted from 40 Gy/20 fractions to 4 Gy/2 fractions, 6 Gy/3 fractions, or 8 Gy/4 fractions. The study aims to evaluate the efficacy and safety of this treatment model, providing further evidence for neoadjuvant treatment strategies in locally advanced esophageal cancer patients.

Additionally, exploratory analyses will be conducted on preoperative and postoperative tissue and blood samples to understand the impact of preoperative low-dose radiotherapy combined with immunotherapy on the immune microenvironment of esophageal cancer, identify appropriate biomarkers, and determine the optimal beneficiary population.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed thoracic esophageal squamous cell carcinoma with clinical staging of: cT1b-cT2 N1-2 M0 or cT3-cT4a N0-2 M0 (AJCC/UICC esophageal cancer staging, 8th edition)
2. Candidates eligible for an R0 curative resection
3. ECOG performance status of 0-1
4. Male or female patients aged ≥18 years and ≤75 years
5. Adequate major organ and bone marrow function (without transfusion or medication correction): Complete blood count: White blood cells ≥ 3.5×10^9/L, Absolute Neutrophil Count (ANC) ≥1.5 ×10^9/L, Platelets ≥100×10^9/L, Hemoglobin ≥9g/dL
6. Radiation oncologist assessment confirms no severe pulmonary ventilatory dysfunction and no acute cardiac failure. (Pulmonary function: FEV1/FVC≥70%, FEV1≥50% of the normal value, DLCO (lung diffusion capacity) actual versus predicted value >80%)
7. Liver function: Total bilirubin ≤1.5 times the upper limit of normal (ULN), Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) ≤2.5 times ULN, Serum albumin ≥3g/dL
8. Renal function: Serum creatinine ≤1.5×ULN, or creatinine clearance ≥ 60ml/min (calculated using the Cockcroft/Gault formula): Female: CrCl = (140 - age) x weight (kg) x 0.85 / 72 x serum creatinine (mg/dL) Male: CrCl = (140 - age) x weight (kg) x 1.00 / 72 x serum creatinine (mg/dL)
9. Study participants voluntarily join the study and sign a written informed consent form, and are able to comply with the protocol-specified visits and related procedures
10. Expected survival >6 months
11. Patients agree to undergo surgical treatment as well as radiotherapy, chemotherapy, and immunotherapy
12. Women of childbearing potential must have a negative pregnancy test within 7 days prior to the initiation of treatment; all participants, regardless of gender, are willing to use appropriate contraceptive methods during the trial and for 8 weeks after the last dose of study medication
13. No esophageal perforation or active esophageal bleeding, and no tracheal or major thoracic vascular invasion
14. According to the solid tumor response evaluation criteria (RECIST version 1.1), at least one measurable lesion by imaging

Exclusion Criteria:

1. Patients who are unsuitable for the immunotherapy and chemotherapy specified in the protocol
2. Patients with a history of treatment for ESCC, including experimental drugs, chemotherapy, radiotherapy, or therapies targeting T-cell co-stimulation checkpoint pathways such as anti-PD-1, anti-PD-L1, anti-PD-L2 antibodies or drugs
3. Patients with a history of primary tumor infiltration causing fistula
4. Patients assessed as having a high risk of fistula or signs of perforation
5. Patients who have required systemic corticosteroid treatment (prednisone > 10 mg/day or equivalent dosage) or other immunosuppressive therapies within 14 days prior to the first administration. However, use of adrenocortical replacement steroids (prednisone ≤ 10 mg/day or equivalent) and minimal systemic absorption of topical, ocular, intra-articular, nasal, and inhaled corticosteroids, as well as short-term (≤ 7 days) use of corticosteroids for non-autoimmune conditions are allowed (dexamethasone can be used for paclitaxel pre-treatment)
6. Patients with active autoimmune diseases or a history of autoimmune diseases that might recur. However, participants with well-controlled type 1 diabetes, hypothyroidism requiring only hormone replacement, well-controlled celiac disease, and non-systemic treated skin conditions like vitiligo, psoriasis, or alopecia, or conditions not likely to recur without an external trigger are eligible
7. Patients with a history of interstitial lung disease, non-infectious pneumonia, or poorly controlled pulmonary diseases including pulmonary fibrosis or acute lung diseases
8. Patients needing systemic antibacterial, antifungal, or antiviral treatment for infections such as tuberculosis. Patients who have had a severe infection including but not limited to hospitalization-required complications, bacteremia, or severe infectious pneumonia within 4 weeks before the first administration, or those who have received therapeutic oral or intravenous antibiotics within 2 weeks before the first administration
9. Patients with a history of allogeneic organ transplant (excluding corneal transplant) or allogeneic hematopoietic stem cell transplant
10. Patients known to be allergic to the study drug tiragolumab, or to the active ingredients or excipients in the combined chemotherapy drugs
11. Patients with significant and severely symptomatic rhythm, conduction, or morphological abnormalities on a resting electrocardiogram, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmias, atrial fibrillation; unstable angina, congestive heart failure, or chronic heart failure with an NYHA classification of ≥ 2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | Immediately after the surgery
  The proportion of subjects with 0% of surviving tumor cells remaining in the primary tumor and in the sampled lymph nodes as evaluated by histology.

SECONDARY OUTCOMES:
Major pathological response | Immediately after the surgery
  Complete response (CR) + partial response (PR) was evaluated by RECIST 1.1 criteria Complete response (CR) + partial response (PR) was evaluated by RECIST 1.1 criteria Complete response (CR) + partial response (PR) was evaluated by RECIST 1.1 criteria
R0 rate | During the surgery
  Intraoperative evaluation
1/2 year event-free survival | 2 years
  The time of enrollment (i.e., signing the ICF) until the following events: any disease progression resulting in surgery not being performed, disease progression or recurrence after surgery, disease progression in patients without surgery, or death from any cause
Overall Response Rate | Immediately after the surgery
  Complete response (CR) + partial response (PR) was evaluated by RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Xue, professor, Principal Investigator — West China Hospital
Locations (1):
- Sichuan University West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klug F, Prakash H, Huber PE, Seibel T, Bender N, Halama N, Pfirschke C, Voss RH, Timke C, Umansky L, Klapproth K, Schakel K, Garbi N, Jager D, Weitz J, Schmitz-Winnenthal H, Hammerling GJ, Beckhove P. Low-dose irradiation programs macrophage differentiation to an iNOS(+)/M1 phenotype that orchestrates effective T cell immunotherapy. Cancer Cell. 2013 Nov 11;24(5):589-602. doi: 10.1016/j.ccr.2013.09.014. Epub 2013 Oct 24. PMID 24209604
- [Background] Herrera FG, Ronet C, Ochoa de Olza M, Barras D, Crespo I, Andreatta M, Corria-Osorio J, Spill A, Benedetti F, Genolet R, Orcurto A, Imbimbo M, Ghisoni E, Navarro Rodrigo B, Berthold DR, Sarivalasis A, Zaman K, Duran R, Dromain C, Prior J, Schaefer N, Bourhis J, Dimopoulou G, Tsourti Z, Messemaker M, Smith T, Warren SE, Foukas P, Rusakiewicz S, Pittet MJ, Zimmermann S, Sempoux C, Dafni U, Harari A, Kandalaft LE, Carmona SJ, Dangaj Laniti D, Irving M, Coukos G. Low-Dose Radiotherapy Reverses Tumor Immune Desertification and Resistance to Immunotherapy. Cancer Discov. 2022 Jan;12(1):108-133. doi: 10.1158/2159-8290.CD-21-0003. Epub 2021 Sep 3. PMID 34479871
- [Background] Gupta A, Probst HC, Vuong V, Landshammer A, Muth S, Yagita H, Schwendener R, Pruschy M, Knuth A, van den Broek M. Radiotherapy promotes tumor-specific effector CD8+ T cells via dendritic cell activation. J Immunol. 2012 Jul 15;189(2):558-66. doi: 10.4049/jimmunol.1200563. Epub 2012 Jun 8. PMID 22685313
- [Background] Barsoumian HB, Ramapriyan R, Younes AI, Caetano MS, Menon H, Comeaux NI, Cushman TR, Schoenhals JE, Cadena AP, Reilly TP, Chen D, Masrorpour F, Li A, Hong DS, Diab A, Nguyen QN, Glitza I, Ferrarotto R, Chun SG, Cortez MA, Welsh J. Low-dose radiation treatment enhances systemic antitumor immune responses by overcoming the inhibitory stroma. J Immunother Cancer. 2020 Oct;8(2):e000537. doi: 10.1136/jitc-2020-000537. PMID 33106386

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT06446726/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT06446726/ICF_001.pdf